CLINICAL TRIAL: NCT05576181
Title: A Single Dose-escalation Study to Evaluate the Safety and Efficacy of Allogeneic CAR-T Targeting CD19 Bridging Hematopoietic Stem Cell Transplantation in Patients With Refractory or Relapsed B Cell Acute Lymphoblastic Leukemia
Brief Title: Safety and Efficacy of ThisCART19A Bridging Hematopoietic Stem Cell Transplantation in Patients With Refractory or Relapsed B-cell Acute Lymphoblastic Leukemia
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundamenta Therapeutics, Ltd. (Industry)
Collaborators: The First Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ThisCART19 FT400-007
Record Dates: First submitted 2022-09-23; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-09

CONDITIONS: Allogeneic, CAR-T, Protein Sequestration, Non-gene Edited
MeSH Terms: interventions — fludarabine; Cyclophosphamide; Etoposide

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ThisCART19A cells infusion and HSCT (Experimental): In this study, allogeneic anti-CD19 CAR T cell (ThisCART19A) infusion is used to treat patients with refractory or relapsed CD19 positive B cell acute lymphoblastic leukemia.
  After patients achieve MRD- remissions through ThisCART19A, they will subsequently receive hematological stem cell transplantations.
  Interventions: Drug: ThisCART19A; Drug: Fludarabine Oral Tablet; Drug: Cyclophosphamide; Drug: VP-16; Procedure: HSCT

INTERVENTIONS:
Drug: ThisCART19A — ThisCART19A is a new type CAR-T therapy for patients with r/r B-ALL.
Drug: Fludarabine Oral Tablet — Fludarabine is used for lymphodepletion.
Drug: Cyclophosphamide — Cyclophosphamide is used for lymphodepletion.
Drug: VP-16 — VP-16 is used for lymphodepletion.
  Other Names: etoposide
Procedure: HSCT — Hematological stem cell transplantation

SUMMARY:
This is a a phase 1, open label study to assess the safety and efficacy of ThisCART19 (Allogeneic CAR-T targeting CD19) Bridging Hematopoietic Stem Cell Transplantation in patients with refractory or relapsed B cell acute lymphoblastic leukemia (r/r B-ALL).

DETAILED DESCRIPTION:
This is a phase 1, single-center, nonrandomized, open-label, dose-escalation study to evaluate the safety and efficacy of ThisCART19A Bridging Hematopoietic Stem Cell Transplantation in patients with CD19 positive r/r B-ALL and identify a treatment regimen most likely to result in clinical efficacy while maintaining a favorable safety profile.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects or legal representatives must sign a voluntary letter of consent approved by the IRB in person prior to the commencement of any screening procedure;
2. Patients diagnosed with B-ALL;
3. No gender limitation, Age 14 years to 75 years (both upper and lower limits included);
4. Consistent with the diagnosis of recurrent refractory B-ALL. Recurrence： was defined as the recurrence of lymphoblasts（≥5%） in peripheral blood or bone marrow or extramedullary diseasefor patients who had acquired CR ; Refractory ：was defined as failure to CR or CRi at the end of induction therapy (generally referred to 4-week regimen or Hyper-CVAD regimen);Patients with Ph+ R/R ALL who failed after 2-line TKI treatment, were intolerant to TKI treatment or were not suitable for TKI treatment; The following factors can coexist:

   1. Failure to prepare autologous CAR-T (definition: too few autologous lymphocytes [200/ML] or cannot meet the release standard);
   2. Experienced treatment with auto car-T/berintoomumab/ CD22 antibody conjugation drugs;
   3. ≥100 days after hematopoietic stem cell transplantation;
   4. High-risk patients (High risk was defined as a high white blood cell count ≥30×109/L at diagnosis or with poor cytogenetic prognosis);

      * Hypodiploid (<44 chromosomes);
      * KMT2A rearrangement: t (4;11) or otherwise;
      * t (v; 14q32) /IgH
      * t (9; 22) (q34; q11.2) or BCR-ABL1
      * Complex karyotype (≥5 chromosomal abnormalities);
      * BCR-ABL1-like (Ph-like) ALL;
      * JAK-STAT (CRLF2r, EPORr, JAK1/2/3r, TYK2r, mutations of SH2B3, IL7r, Jak1/2/3);
      * ABL class rearrangements (such as ABL1, ABL2, PDGFRA, PDGFRB, FGFR, etc.)
      * Others (NTRKr, FLT3r, LYNr, PTK2Br);
      * Intrachromosomal amplification of chromosome 21 (iAMP21);
      * t (17; 19): TCF3-HLF fusion;
      * Alterations of IKZF1;
   5. Extramedullary lesions.
5. The expected survival time is ≥12 weeks;
6. ECOG score 0-2;
7. Adequate bone marrow, renal, hepatic, pulmonary and cardiac function;
8. CD19 was still expressed in leukemia cells in bone marrow, peripheral blood or biopsy tissue by flow cytometry within one month prior to informed consent (after the last treatment).

Exclusion Criteria:

1. Allergic to preconditioning measures;
2. Diagnosis of chronic myelogenous leukemia lymphoid blast crisis;
3. Isolated extramedullary relapse;
4. Presence of CNS-3 disease or CNS-2 disease with neurological changes;
5. Imaging confirmed the presence of central nervous system involvement;
6. Severe CNS disorders such as a history of frequent epileptic seizures;
7. Patients with other malignancies other than B-cell malignancies within 5 years prior to screening. Patients with cured skin squamous carcinoma, basal carcinoma, non-primary invasive bladder cancer, localized low-risk prostate cancer, in situ cervical/breast cancer can be recruited.
8. Uncontrollable bacterial, fungal and viral infection during screening;
9. Patients had pulmonary embolism (PE) and/or deep vein thrombosis (DVT) within 3 months prior to enrollment;
10. Had intolerant severe cardiovascular and cerebrovascular diseases and hereditary diseases prior to enrollment;
11. Radiation therapy within 2 weeks prior to lymphodepletion chemotherapy (>30% bone marrow exposure);
12. Active hepatitis B virus (HBV) or hepatitis C virus (HCV) or Human immunodeficiency virus (HIV) or Syphilis infection. HBV-DNA < 2000 IU/mL can be enrolled, but should admitted to use anti-virus drugs such as entecavir, tenofovir, etc, and supervisory the relative indication during the treatment;
13. Vaccinated with influenza vaccine within 2 weeks prior to lymphodepleting chemotherapy (Severe Acute Respiratory Syndrome-Corona virus disease 19 can be included, inactivated, live/non-live adjuvant vaccinations allowed to be included) ;
14. Patients who are receiving Graft versus host disease Hepatitis(GvHD) treatment; Patients without GvHD and who had stopped immunosuppressive drugs for at least 1 month were eligible for inclusion;
15. Women who are in pregnant or lactating, and female subjects or partners who plan to be pregnant within 1 year after cell infusion. Male subjects who plan pregnancy within 1 year after infusion;
16. Any ineligibility conditions considered by the investigator that may increase the risk of the subject or interfere with the results of the study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 19 (Estimated)
Dates: Start 2022-10-15 (Estimated); Primary Completion 2025-01-22 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) observation in patient with B-ALL in each dose level during dose escalation and dose expansion stage | 28 days
  DLT is defined as the incidence of severe adverse events related to ThisCART19A more than 33% in each dose level.
Overall Complete Response (OCR) Rate (Complete Remission [CR]+ Complete Remission With Incomplete Hematologic Recovery [CRi]) within 3 months | 3 months
  OCR rate within 3 months: percentage of participants achieving CR+CRi within 3 months after CAR-T cell infusion.

SECONDARY OUTCOMES:
Minimum Residual Disease (MRD) Negative Remission Rate | 3 months
  MRD was assessed utilizing multicolor flow cytometry to detect residual cancerous cells with a sensitivity of 10^-4. MRD negative remission was defined as MRD < 10^-4 threshold. Percentage of participants with MRD negative remission was reported.
Duration of response(DOR) during dose escalation stage and expansion stage | 24 months
  DOR was defined as the time from first CR or CRi to relapse or any death in the absence of documented relapse.
RFS (Relapse-free Survival) | 24 months
  RFS is defined as the time from the date of ThisCART19A infusion to the date of disease relapse or death from any cause.
EFS (Event-free Survival) | 24 months
  EFS is defined as the time from the date of ThisCART19A infusion to the date of disease relapse, progression, genetic relapse or death from any cause.
OS (Overall Survival) | 24 months
  OS is defined as the time from the date of ThisCART19A infusion to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Ph.D, Principal Investigator — The First Affiliated Hospital of Zhengzhou University

IPD SHARING:
Plan to Share IPD: No